CLINICAL TRIAL: NCT02636439
Title: Study of the Effects Caloric Restriction and Exercise Training in Patients With Heart Failure and a Normal Ejection Fraction
Brief Title: Exercise Intolerance in Elderly Patients With HFpEF(Heart Failure With Preserved Ejection Fraction)
Acronym: SECRET-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00032364; R01AG018915 (NIH)
Record Dates: First submitted 2015-12-09; First posted 2015-12-21 (Estimated); Results first posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2020-12

CONDITIONS: Heart Failure, Diastolic; Obesity
Keywords: Diastolic heart failure; Heart Failure; Elderly; Obesity
MeSH Terms: conditions — Heart Failure, Diastolic; Obesity; Heart Failure | interventions — Diet; Resistance Training; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dietary, and aerobic exercise (Active Comparator): Intervention for diet-A hypocaloric diet will be developed to achieve a 2800 kcal/week deficit, which should produce about 0.4 kg (1 lb.) weight loss per week.
  Intervention for aerobic exercise-Based on initial evaluations and the stress testing results, (HR, VO2, RPE) an individual exercise prescription will be developed for aerobic training.
  Interventions: Behavioral: dietary, and aerobic exercise
- dietary, aerobic and resistance training (Active Comparator): Intervention for diet-A hypocaloric diet will be developed to achieve a 2800 kcal/week deficit, which should produce about 0.4 kg (1 lb.) weight loss per week.
  Intervention for aerobic exercise-Based on initial evaluations and the stress testing results, (HR, VO2, RPE) an individual exercise prescription will be developed for aerobic training.
  Intervention for resistance training- Additional weight resistant exercise will be added to this arm.
  Interventions: Behavioral: dietary, aerobic and resistance training; Behavioral: dietary, and aerobic exercise

INTERVENTIONS:
Behavioral: dietary, aerobic and resistance training — hypocaloric diet individual exercise prescription for aerobic training individual exercise prescription for resistance training.
  Arms: dietary, aerobic and resistance training
Behavioral: dietary, and aerobic exercise — hypocaloric diet individual prescription for aerobic training.

SUMMARY:
The purpose of this study is to examine the effects of weight loss via hypocaloric diet (CR)and aerobic exercise (AT) compared to the effects of weight loss via hypocaloric diet (CR), aerobic training (AT)and resistance training (RT).

DETAILED DESCRIPTION:
Heart failure with preserved ejection fraction (HFPEF) is the most common form of HF, is nearly unique to the older population, particularly older women, and is increasing in prevalence. Exercise intolerance, with severe exertional dyspnea and fatigue, is the primary manifestation of chronic HFPEF and is a major determinant of these patients' severely reduced quality of life (QOL). However, its pathophysiology is poorly understood and its optimal treatment remains undefined.

Our recent data and others' indicate that in older HFPEF patients, both increased adiposity and abnormalities in skeletal muscle are major contributors to exercise intolerance and potential therapeutic targets. Obesity is one of the strongest risk factors for HFPEF, and is a robust predictor of physical disability in older persons. The investigator recently reported that in HFPEF compared to age-matched controls, percent total and leg lean mass are significantly reduced and independently predict exercise capacity.

Using MRI and needle biopsy of the thigh muscle, the investigators found increased fat infiltration, reduced capillary density and percent type I oxidative fibers, and trends for reduced muscle mitochondrial mass and function. Reduced exercise capacity was related to each of these muscle abnormalities, supporting their important role in HFPEF.

Diet, with or without aerobic exercise, can increase exercise capacity and quality of life in older obese persons with a variety of disorders, but usually results in significant loss of skeletal muscle mass, which could potentially have adverse long term consequences. The purpose of this trial is to determine if addition of resistance training to diet plus aerobic exercise training can improve skeletal muscle mass and function in HFPEF.

Multiple lines of evidence and our preliminary data indicate that resistance training (RT) may be an ideal addition to CR+AT for HFPEF, since RT reliably increases muscle mass, quality, strength, and function, significantly more than AT, and can prevent nearly 50% of the muscle mass loss during CR.

Therefore, the primary aim of the proposed study is to conduct a randomized, single-blinded 20-week intervention trial of RT added to CR+AT in 84 overweight / obese (BMI greater than 28 kg/m2), older (age greater than 60 years) HFPEF patients to test the following primary hypothesis:

The addition of resistance training to CR+AT will improve exercise capacity.

ELIGIBILITY:
Inclusion Criteria:

1. Age 60 years or older
2. Ejection fraction ≥ 50%
3. Left Ventricular Diastolic Dysfunction ≥ grade 1
4. BMI ≥ 28 kg/m2
5. HF symptoms/ signs by cardiologist review, using NHANES HF Clinical Score >/= 3 or Rich et al. criteria for HF

Exclusion Criteria:

1. Valvular heart disease as the primary etiology of CHF (congestive heart failure)
2. Significant change in cardiac medication or Heart Failure symptoms <6 weeks
3. Hospitalization or urgent care visit <6 weeks
4. Uncontrolled hypertension
5. Uncontrolled diabetes
6. Evidence of significant Chronic Obstructive Pulmonary Disease (COPD)
7. Recent or debilitating stroke
8. Cancer or other noncardiovascular conditions with life expectancy less than 2 years
9. Significant anemia (<10 g/dL Hgb)
10. Significant renal insufficiency (eGFR <30 mL/min/1.73m2)
11. Pregnant or of child-bearing potential
12. Psychiatric disease- uncontrolled major psychoses, depressions, dementia, or personality disorder
13. Plans to leave area within the study period
14. Refuses informed consent -

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dalane W Kitzman, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schaich CL, Hughes TM, Kitzman DW, Jung Y, Chen H, Nicklas BJ, Houston DK, Brubaker PH, Molina AJA, Hugenschmidt CE. Neurocognitive Impairments and Their Improvement Following Exercise and Dietary Interventions in Older Patients With Heart Failure With Preserved Ejection Fraction. Circ Heart Fail. 2024 Jan;17(1):e011134. doi: 10.1161/CIRCHEARTFAILURE.123.011134. Epub 2023 Dec 1. No abstract available. PMID 38037817
- [Derived] Brubaker PH, Nicklas BJ, Houston DK, Hundley WG, Chen H, Molina AJA, Lyles WM, Nelson B, Upadhya B, Newland R, Kitzman DW. A Randomized, Controlled Trial of Resistance Training Added to Caloric Restriction Plus Aerobic Exercise Training in Obese Heart Failure With Preserved Ejection Fraction. Circ Heart Fail. 2023 Feb;16(2):e010161. doi: 10.1161/CIRCHEARTFAILURE.122.010161. Epub 2022 Oct 31. PMID 36314122

RESULTS

PARTICIPANT FLOW:
Groups:
- Dietary, and Aerobic Exercise: Intervention for diet-A hypocaloric diet will be developed to achieve a 2800 kcal/week deficit, which should produce about 0.4 kg (1 lb.) weight loss per week.
  Intervention for aerobic exercise-Based on initial evaluations and the stress testing results, (HR, VO2, RPE) an individual exercise prescription will be developed for aerobic training.
  dietary, and aerobic exercise: hypocaloric diet individual prescription for aerobic training.
- Dietary, Aerobic, and Resistance Training: Intervention for diet-A hypocaloric diet will be developed to achieve a 2800 kcal/week deficit, which should produce about 0.4 kg (1 lb.) weight loss per week.
  Intervention for aerobic exercise-Based on initial evaluations and the stress testing results, (HR, VO2, RPE) an individual exercise prescription will be developed for aerobic training.
  Intervention for resistance training- Additional weight resistant exercise will be added to this arm.
  dietary, aerobic and resistance training: hypocaloric diet individual exercise prescription for aerobic training individual exercise prescription for resistance training.
  dietary, and aerobic exercise: hypocaloric diet individual prescription for aerobic training.
Period: Overall Study
Arm/Group | Dietary, and Aerobic Exercise | Dietary, Aerobic, and Resistance Training
Started | 44 | 44
Completed | 38 | 41
Not Completed | 6 | 3
Not completed — Adverse Event | 2 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Non-compliance | 1 | 1
Not completed — Personal reasons | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dietary, Aerobic and Resistance Training: Intervention for diet-A hypocaloric diet will be developed to achieve a 2800 kcal/week deficit, which should produce about 0.4 kg (1 lb.) weight loss per week.
  Intervention for aerobic exercise-Based on initial evaluations and the stress testing results, (HR, VO2, RPE) an individual exercise prescription will be developed for aerobic training.
  Intervention for resistance training- Additional weight resistant exercise will be added to this arm.
  dietary, aerobic and resistance training: hypocaloric diet individual exercise prescription for aerobic training individual exercise prescription for resistance training.
  dietary, and aerobic exercise: hypocaloric diet individual prescription for aerobic training.
- Total: Total of all reporting groups
Arm/Group | Dietary, and Aerobic Exercise | Dietary, Aerobic and Resistance Training | Total
Number analyzed (Participants) | 44 | 44 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (5.4) | 69.7 (5.8) | 68.8 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 38 | 75
  Male | 7 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 44 | 44 | 88
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 24 | 23 | 47
  White | 19 | 20 | 39
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 44 | 44 | 88
Peak exercise oxygen consumption (VO2) [Mean (Standard Deviation); unit: ml/min] — Peak exercise oxygen consumption (VO2) assessed during cardiopulmonary exercise test using expired gas analysis.
  ml/min | 1529 (375) | 1530 (366) | 1530 (368)

OUTCOME MEASURES:

1. Primary Outcome: Peak Exercise Oxygen Consumption (VO2)
Description: Peak exercise oxygen consumption (VO2) pre and post intervention
Time Frame: 20 weeks
Population: Analysis completed on all participants with peak VO2 obtained (n=77).
Measure: Least Squares Mean (Standard Error); unit: ml/min
Arm/Group | Dietary, and Aerobic Exercise | Dietary, Aerobic, and Resistance Training
Number analyzed (Participants) | 38 | 39
ml/min | 1609 (24) | 1653 (24)
Statistical Analysis 1: Comparison: Dietary, and Aerobic Exercise vs Dietary, Aerobic, and Resistance Training; Test type: Superiority; p = 0.21, ANCOVA; adjusted for baseline value, age, and sex; Mean Difference (Final Values) = 44, 95% CI 2-sided [-25 to 112]

2. Secondary Outcome: Skeletal Muscle Mass
Description: Measure skeletal muscle mass in kg by DEXA analysis pre and post intervention.
Time Frame: 20 weeks
Population: Analysis completed on all participants with DEXA measurement (n=78).
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Dietary, and Aerobic Exercise | Dietary, Aerobic, and Resistance Training
Number analyzed (Participants) | 38 | 40
kg | 49.4 (0.3) | 49.4 (0.3)
Statistical Analysis 1: Comparison: Dietary, and Aerobic Exercise vs Dietary, Aerobic, and Resistance Training; Test type: Superiority; p = 0.86, ANCOVA; Adjusted for baseline value, age, and sex; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-1.0 to 0.8]

3. Secondary Outcome: Thigh Skeletal Muscle Mass
Description: Measure skeletal muscle mass by MRI analysis pre and post intervention.
Time Frame: 20 weeks
Population: Analysis completed on all participants with thigh MRI.
Measure: Least Squares Mean (Standard Error); unit: cm^2
Arm/Group | Dietary, and Aerobic Exercise | Dietary, Aerobic, and Resistance Training
Number analyzed (Participants) | 39 | 40
cm^2 | 108.5 (1.2) | 108.9 (1.1)
Statistical Analysis 1: Comparison: Dietary, and Aerobic Exercise vs Dietary, Aerobic, and Resistance Training; Test type: Superiority; p = 0.77, ANCOVA; Adjusted for baseline value, age, and sex; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-2.8 to 3.8]

4. Secondary Outcome: Thigh Muscle Composition
Description: MRI skeletal muscle to intermuscular fat ratio
Time Frame: 20 weeks
Population: Analysis completed on all participants with MRI measurements.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Dietary, and Aerobic Exercise | Dietary, Aerobic, and Resistance Training
Number analyzed (Participants) | 39 | 40
ratio | 4.0 (0.1) | 4.0 (0.1)
Statistical Analysis 1: Comparison: Dietary, and Aerobic Exercise vs Dietary, Aerobic, and Resistance Training; Test type: Superiority; p = 0.85, ANCOVA; Adjusted for baseline value, age, and sex; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.3 to 0.2]

5. Secondary Outcome: Muscle Strength
Description: maximal isokinetic knee extensor strength (Newton-meters, Nm) using an isokinetic dynamometer (Biodex®)
Time Frame: 20 weeks
Population: Analysis completed on all participants with Biodex measures.
Measure: Least Squares Mean (Standard Error); unit: Nm
Arm/Group | Dietary, and Aerobic Exercise | Dietary, Aerobic, and Resistance Training
Number analyzed (Participants) | 25 | 28
Nm | 97.5 (2.3) | 103.9 (2.2)
Statistical Analysis 1: Comparison: Dietary, and Aerobic Exercise vs Dietary, Aerobic, and Resistance Training; Test type: Superiority; p = 0.053, ANCOVA; Adjusted for baseline value, age, and sex; Mean Difference (Final Values) = 6.4, 95% CI 2-sided [-0.1 to 12.9]

6. Secondary Outcome: Muscle Quality
Description: knee extensor strength to thigh muscle area assessed by MRI (Nm/cm2).
Time Frame: 20 weeks
Population: Analysis completed on all participants with MRI and Biodex measurements.
Measure: Least Squares Mean (Standard Error); unit: Nm/cm^2
Arm/Group | Dietary, and Aerobic Exercise | Dietary, Aerobic, and Resistance Training
Number analyzed (Participants) | 25 | 27
Nm/cm^2 | 0.90 (0.02) | 0.97 (0.02)
Statistical Analysis 1: Comparison: Dietary, and Aerobic Exercise vs Dietary, Aerobic, and Resistance Training; Test type: Superiority; p = 0.043, ANCOVA; Adjusted for baseline value, age, and sex; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [0.00 to 0.13]

7. Secondary Outcome: Quality of Life Measured by Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Summary Score
Description: The KCCQ Overall Summary Summary Score is a heart failure disease-specific quality of life measure encompassing domains of physical limitation, HF symptoms, quality of life, and social limitation scored on a scale of 0-100 with higher scores indicating better health status.
Time Frame: 20 weeks
Population: Analysis completed on all participants with KCCQ assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Dietary, and Aerobic Exercise | Dietary, Aerobic, and Resistance Training
Number analyzed (Participants) | 38 | 41
score on a scale | 91 (2) | 87 (2)
Statistical Analysis 1: Comparison: Dietary, and Aerobic Exercise; Test type: Superiority; p = 0.07, ANCOVA; Adjusted for baseline value, age, and sex; Mean Difference (Final Values) = -5, 95% CI 2-sided [-10 to 0]

8. Secondary Outcome: Quality of Life Measured by Short Form 36 Item Questionnaire (SF-36)
Description: The SF-36 is a quality of life assessment with 2 component scores (Physical Composite Score and Mental Composite Score) ranging 0-100 with higher scores indicating better health status.
Time Frame: 20 weeks
Population: Analysis completed on all participants with SF-36 assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Dietary, and Aerobic Exercise | Dietary, Aerobic, and Resistance Training
Number analyzed (Participants) | 37 | 40
score on a scale | 47.4 (1.4) | 46.9 (1.3)
Statistical Analysis 1: Comparison: Dietary, and Aerobic Exercise vs Dietary, Aerobic, and Resistance Training; Test type: Superiority; p = 0.79, ANCOVA; Adjusted for baseline value, age, and sex; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-4.4 to 3.3]

9. Other Pre Specified Outcome: Mitochondrial Content
Description: Porin citrate synthase pre and post intervention.
Time Frame: 20 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Mitochondrial Function
Description: respiratory control ratio and mitofusin 2 concentration.pre and post intervention.
Time Frame: 20 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 20 weeks
Arm/Group | Dietary, and Aerobic Exercise | Dietary, Aerobic, and Resistance Training
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 6/44 | 6/44
Other Adverse Events (participants affected / at risk) | 24/44 | 25/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dietary, and Aerobic Exercise (N=44) | Dietary, Aerobic, and Resistance Training (N=44)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Heart failure exacerbation (Cardiac disorders) | 0 (0) | 1 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Atypical chest pain (General disorders) | 1 (1) | 0 (0)
Rectal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Spinal surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dietary, and Aerobic Exercise (N=44) | Dietary, Aerobic, and Resistance Training (N=44)
Abscess (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
acute pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 3 (3)
bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
broken tooth (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
chest pain (Cardiac disorders) | 2 (3) | 3 (3)
heart failure exacerbation (Cardiac disorders) | 1 (1) | 1 (1)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
elevated ocular pressure (Eye disorders) | 0 (0) | 1 (1)
esophageal spasm (Gastrointestinal disorders) | 1 (1) | 0 (0)
fall (Injury, poisoning and procedural complications) | 6 (7) | 6 (7)
foot pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 1 (1) | 0 (0)
hypertension (Vascular disorders) | 1 (1) | 0 (0)
hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
hypotension (Vascular disorders) | 0 (0) | 1 (1)
knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (7)
finger laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
muscle strain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
post-menopausal bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
presyncope (Nervous system disorders) | 4 (4) | 0 (0)
shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
upper respiratory infection (Infections and infestations) | 1 (1) | 1 (2)
urinary tract infections (Renal and urinary disorders) | 0 (0) | 2 (2)
vomitting (Gastrointestinal disorders) | 2 (2) | 0 (0)
dizziness (Nervous system disorders) | 1 (1) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
hip pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-02): https://cdn.clinicaltrials.gov/large-docs/39/NCT02636439/Prot_SAP_001.pdf
  • Informed Consent Form (2019-05-31): https://cdn.clinicaltrials.gov/large-docs/39/NCT02636439/ICF_000.pdf